CLINICAL TRIAL: NCT04107922
Title: Metabolic Actions of a Supplement of Ilex Paraguariensis, White Mulberry and Chromium Picolinate in Non-diabetic Subjects With Dysglycemia, a Randomized Clinical Trial
Brief Title: Nutraceutical on Hyperglycemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Giuseppe Derosa, MD, PhD, FESC, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: P-20180016364
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Dysglycemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glicoset (Active Comparator): Glicoset is a nutraceutical containing Ilex Paraguariensis, White Mulberry and Chromium Picolinate
  Interventions: Dietary Supplement: Glicoset
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Glicoset — Patients will take a nutraceutical containing Ilex Paraguariensis, White Mulberry and Chromium Picolinate
  Arms: Glicoset
Other: Placebo — Patients will take placebo
  Arms: Placebo

SUMMARY:
The aim will be to evaluate if Glicoset® 1000, a nutraceutical containing Ilex Paraguariensis, White Mulberry and Chromium Picolinate, can be effective in improving glycemic status in subject with dysglycemia.

DETAILED DESCRIPTION:
The aim will be to evaluate if Glicoset® 1000, a nutraceutical containing Ilex Paraguariensis, White Mulberry and Chromium Picolinate, can be effective in improving glycemic status in subject with dysglycemia.

The investigators will enroll patients with impaired fasting plasma glucose (IFG) or impaired glucose tolerance (IGT), not taking hypoglycemic agents (both pharmaceuticals or nutraceutical agents). Patients will be randomized to take placebo or Glicoset® 1000 for 3 months, in a randomized, double-blind, placebo-controlled design. Glicoset® 1000 and placebo will be self-administered once a day, 1 tablet during the breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Patients with impaired fasting glucose (IFG) or impaired fasting glucose (IGT)
* Patients not taking hypoglycemic agents (both pharmaceuticals or nutraceutical agents)

Exclusion Criteria:

* Patients with type 1 or type 2 diabetes mellitus
* Patients with impaired hepatic function
* Patient with impaired renal function
* Patients with gastrointestinal disorders
* Patients with current or previous evidence of ischemic heart disease, heart failure, or stroke
* Patients with weight change of > 3 Kg during the preceding 3 months
* Patients with hystory of malignancy, and significant neurological or psychiatric disturbances, including alcohol or drug abuse.
* Patients taking (within the previous 3 months) hypoglycemic agents, laxatives, beta-agonists (other than inhalers), cyproheptadine, anti-depressants, antiserotoninergics, phenothiazines, barbiturates, oral corticosteroids, and antipsychotics
* Women who were pregnant or breastfeeding or of childbearing potential and not taking adequate contraceptive precautions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Progression of dysglicemia | 3 months
  Oral glucose tolerance test

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Matteo, Pavia, Lombardy, Italy